CLINICAL TRIAL: NCT05710510
Title: Rural Engagement in TelemedTeam for Options in Obesity Treatment Solutions (RE-TOOL)
Brief Title: Rural Engagement in TelemedTeam for Options in Obesity Treatment Solutions
Acronym: RE-TOOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00147574; 1R01CA268034-01 (NIH)
Record Dates: First submitted 2022-12-29; First posted 2023-02-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Weight loss; Weight management; Behavioral intervention; Medical management of obesity; Team care
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss | interventions — Models, Biological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Care + Model (Active Comparator): Quarterly clinic visits with a local primary care provider
  Interventions: Behavioral: Local Care + Model
- Team Care Model (Active Comparator): An intensive group lifestyle intervention led by a lifestyle coach via Zoom, paired with quarterly clinic visits with a local primary care provider and the lifestyle coach, the coach joining via telemedicine.
  Interventions: Behavioral: Team Care Model

INTERVENTIONS:
Behavioral: Local Care + Model — Local primary care providers receive training in medical management of obesity prior to the start of the participant intervention.
  Participants receive 6 quarterly clinic visits with their local primary care provider focused on medical management of obesity.
  Arms: Local Care + Model
Behavioral: Team Care Model — Local primary care providers receive training in medical management of obesity prior to the start of the participant intervention.
  Participants receive an intensive 18-month group lifestyle intervention (30 total sessions) led by a study lifestyle coach via Zoom, and 6 quarterly 1:1 visits via Zoom with their lifestyle coach. Participants also receive 6 quarterly clinic visits with their local primary care provider; the study lifestyle coach joins the visits via telemedicine. All three parties may meet via telemedicine if needed. The group lifestyle intervention is led by obesity treatment specialists with relevant graduate training and experience.
  Arms: Team Care Model

SUMMARY:
The purpose of this study is to compare two methods for managing obesity in rural primary care patients. The first method includes quarterly 1:1 meetings with the participant and their primary care provider and the second includes a group lifestyle intervention over Zoom paired with quarterly team meetings with the participant, their primary care provider and their lifestyle coach, the coach joining via Zoom. Investigators will evaluate which method is best at helping participants lose weight over 18 months.

DETAILED DESCRIPTION:
Obesity increases risk for 13 types of cancer and now affects over 40% of the U.S. adult population, with even higher prevalence among rural Americans. Rural residents often lack access to weight control programs and food and physical activity resources that promote healthy lifestyles, especially in small or remote rural areas. It is important for obesity treatment to be offered in rural primary care, yet local resources are often lacking. Medical management by a primary care provider (PCP) during behavioral weight loss is essential to address co-morbid medical conditions, evaluate obesogenic medications, and explore options for guideline-recommended pharmacotherapy and surgical treatment. This study is designed to enhance sustainable access to obesity treatment in rural communities by offering education to local providers on obesity management and integrating team-based care into an obesity treatment model through telemedicine.

The two methods of obesity treatment to be studied are:

* Local Care + Arm: Quarterly clinic visits with the participants and their local primary care provider
* Team Care Arm: An intensive group lifestyle intervention offered by a lifestyle coach via Zoom, paired with quarterly clinic visits with the participant, their local primary care provider and the lifestyle coach, the coach joining via telemedicine.

Participants will be in the study about 18 months. Participants in the Local Care + arm will be asked to complete 4 data collection visits and 6 quarterly clinic visits. Participants in the Team Care arm will be asked to complete 4 data collection visits, 30 counseling sessions and 6 quarterly clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI: >= 30 kg/m2
* Rural resident
* English speaking
* Physician clearance to participate
* Able to walk without assistance
* Seen at least once in their primary care clinic within the past year
* Internet access or smart phone (to access smart scale for weight measurement)

Exclusion Criteria:

* History of myocardial infarction within last six months
* History of stroke within last six months
* History of new cancer diagnosis within last six months
* History of bariatric surgery within the last two years
* Pregnancy within last 6 months or planned within the next 18 months
* Currently breastfeeding
* End stage renal disease, currently on dialysis, or anticipated dialysis or renal transplant within the next 18 months
* End stage liver disease, or anticipated liver transplant within the next 18 months
* Currently enrolled or planning to enroll in another study where weight loss is targeted or weight fluctuation is expected
* Currently planning to move outside of current provider area, or leave primary care clinic within the next 18 months
* Another household member is already participating in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Percent weight loss at 18 months | 18 months
  Mean percent weight loss at 18 months; unadjusted

SECONDARY OUTCOMES:
Percent weight loss at 6 months | 6 months
  Mean percent weight loss at 6 months; unadjusted
Percent weight loss at 12 months | 12 months
  Mean percent weight loss at 12 months; unadjusted
Weight loss (kg) at 6 months | 6 months
  Mean weight loss (kg) at 6 months; unadjusted
Weight loss (kg) at 12 months | 12 months
  Mean weight loss (kg) at 12 months; unadjusted
Weight loss (kg) at 18 months | 18 months
  Mean weight loss (kg) at 18 months; unadjusted
Proportion achieving ≥5% weight loss at 6 months | 6 months
  Proportion achieving ≥5% weight loss at 6 months; unadjusted
Proportion achieving ≥5% weight loss at 12 months | 12 months
  Proportion achieving ≥5% weight loss at 12 months; unadjusted
Proportion achieving ≥5% weight loss at 18 months | 18 months
  Proportion achieving ≥5% weight loss at 18 months; unadjusted
Proportion achieving ≥10% weight loss at 6 months | 6 months
  Proportion achieving ≥10% weight loss at 6 months; unadjusted
Proportion achieving ≥10% weight loss at 12 months | 12 months
  Proportion achieving ≥10% weight loss at 12 months; unadjusted
Proportion achieving ≥10% weight loss at 18 months | 18 months
  Proportion achieving ≥10% weight loss at 18 months; unadjusted
Change in diet quality at 6 months | Baseline and 6 months
  Mean change in diet quality, measured by Rapid Eating Assessment for Participant--Shortened Version (REAPS) at 6 months; unadjusted. The REAPS estimates diet quality through 13 items which assess weekly eating habits. Possible scores range from 13 (worst diet quality) to 39 (best diet quality).
Change in diet quality at 12 months | Baseline and 12 months
  Mean change in diet quality, measured by Rapid Eating Assessment for Participant--Shortened Version (REAPS) at 12 months; unadjusted. The REAPS estimates diet quality through 13 items which assess weekly eating habits. Possible scores range from 13 (worst diet quality) to 39 (best diet quality).
Change in diet quality at 18 months | Baseline and 18 months
  Mean change in diet quality, measured by Rapid Eating Assessment for Participant--Shortened Version (REAPS) at 18 months; unadjusted. The REAPS estimates diet quality through 13 items which assess weekly eating habits. Possible scores range from 13 (worst diet quality) to 39 (best diet quality).
Change in physical activity at 6 months | Baseline and 6 months
  Mean change in MET-HOURS per week measured by Modifiable Activity Questionnaire (MAQ) at 6 months; unadjusted. The MAQ will be used to measure participants' leisure-time physical activity over the past 7 days. Leisure-time physical activity will be calculated as the Metabolic Equivalent of Task (MET) hours per week (MET-hr/week) and estimated by multiplying time (in hours) spent in an activity by the activities estimated MET and summing across all activities.
Change in physical activity at 12 months | Baseline and 12 months
  Mean change in MET-HOURS per week measured by Modifiable Activity Questionnaire (MAQ) at 12 months; unadjusted. The MAQ will be used to measure participants' leisure-time physical activity over the past 7 days. Leisure-time physical activity will be calculated as the Metabolic Equivalent of Task (MET) hours per week (MET-hr/week) and estimated by multiplying time (in hours) spent in an activity by the activities estimated MET and summing across all activities.
Change in physical activity at 18 months | Baseline and 18 months
  Mean change in MET-HOURS per week measured by Modifiable Activity Questionnaire (MAQ) at 18 months; unadjusted. The MAQ will be used to measure participants' leisure-time physical activity over the past 7 days. Leisure-time physical activity will be calculated as the Metabolic Equivalent of Task (MET) hours per week (MET-hr/week) and estimated by multiplying time (in hours) spent in an activity by the activities estimated MET and summing across all activities.
Change in physical quality of life at 6 months | Baseline and 6 months
  Mean change in physical quality of life, measured by SF-12 at 6 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a physical functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in physical quality of life at 12 months | Baseline and 12 months
  Mean change in physical quality of life, measured by SF-12 at 12 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a physical functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in physical quality of life at 18 months | Baseline and 18 months
  Mean change in physical quality of life, measured by SF-12 at 18 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a physical functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in mental quality of life at 6 months | Baseline and 6 months
  Mean change in mental quality of life, measured by SF-12 at 6 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a mental functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in mental quality of life at 12 months | Baseline and 12 months
  Mean change in mental quality of life, measured by SF-12 at 12 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a mental functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in mental quality of life at 18 months | Baseline and 18 months
  Mean change in mental quality of life, measured by SF-12 at 18 months; unadjusted. The Short Form Health Survey (SF-12) is a general quality of life measure with a mental functioning summary score. Scores range from 0 to 100 with higher scores representing better functioning.
Change in weight-related quality of life at 6 months | Baseline and 6 months
  Mean change in total quality of life, measured by Impact of Weight on Quality of Life-Lite (IWQOL-L) at 6 months; unadjusted. The IWQOL-L measure consists of a total score and five subscales--physical function, self-esteem, sexual life, public distress, and work. The total score ranges from 0 to 100 with higher scores indicating better quality of life.
Change in weight-related quality of life at 12 months | Baseline and 12 months
  Mean change in total quality of life, measured by Impact of Weight on Quality of Life-Lite (IWQOL-L) at 12 months; unadjusted. The IWQOL-L measure consists of a total score and five subscales--physical function, self-esteem, sexual life, public distress, and work. The total score ranges from 0 to 100 with higher scores indicating better quality of life.
Change in weight-related quality of life at 18 months | Baseline and 18 months
  Mean change in total quality of life, measured by Impact of Weight on Quality of Life-Lite (IWQOL-L) at 18 months; unadjusted. The IWQOL-L measure consists of a total score and five subscales--physical function, self-esteem, sexual life, public distress, and work. The total score ranges from 0 to 100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christie Befort, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
A clean, de-identified copy of the final dataset will be created within 30 days of primary outcome paper publication. Data will be made available to researchers upon email request to the Principal Investigator. We will convert date of birth to age, and other identifiers (e.g, address, zip code, state) will be removed. Data and associated documentation will be made available to users under a data-sharing agreement that provides for: (1) a commitment to use the data solely for research purposes and to not identify individual participants during use or publication; (2) a commitment to secure the data using appropriate computer technology upon receipt; and (3) a commitment to destroy or return the data to the KU Medical Center after analyses are completed. Data will be saved as SAS or SPSS files and provided to requesters via KUMC's Secure File Transfer service. A copy of our analytic code used to generate our primary outcomes paper(s) will be made available on request in the same fashion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 30 days of publication of the primary outcome paper
Access Criteria: upon email request to the Principal Investigator